CLINICAL TRIAL: NCT01363024
Title: An Open-Label, Multicenter, Phase I Dose-Escalation Trial Evaluating the Safety and Pharmacokinetics of MFGR1877S in Patients With Advanced Solid Tumors
Brief Title: Trial Evaluating the Safety and Pharmacokinetics of MFGR1877S in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MFG4991g; GO27817 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Solid Tumor
Keywords: Solid Cancers
MeSH Terms: interventions — vofatamab

ARMS (1):
- A (Experimental)
  Interventions: Drug: MFGR1877S

INTERVENTIONS:
Drug: MFGR1877S — Intravenous escalating dose

SUMMARY:
This is a multicenter, open-label, dose-escalation study to assess the safety, tolerability and Pharmacokinetics of MGFR1877S.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy >/= 12 weeks
* ECOG performance status of 0 or 1
* Histologic or cytologic documentation of locally advanced, or metastatic solid malignancy that has relapsed after or failed to respond to at least one prior regimen or for which there is no standard therapy
* Evaluable or measurable disease. Prostate cancer patients with non-measurable disease are eligible if they have two rising prostate-specific antigen (PSA) levels (5 ng/mL measured 2 weeks apart) that meet the PSA Working Group criteria for progression prior to initiation of study treatment. Ovarian cancer patients with non-measurable disease are eligible if they have two rising CA-125 levels greater than the ULN (2 weeks apart prior to initiation of study treatment).
* Adequate hematologic and end organ function
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use an effective form of contraception and to continue its use until 90 days after the last dose of study treatment
* Consent to provide archival tissue

Exclusion Criteria:

* Prior use of any monoclonal antibody within 4 weeks before Cycle 1, Day 1
* Experimental therapy within 4 weeks prior to Cycle 1, Day 1
* Palliative radiotherapy within 2 weeks prior to Cycle 1, Day 1
* Prior anti-cancer therapy within 4 weeks prior to Cycle 1, Day 1
* Major surgical procedure or trauma within 4 weeks prior to Cycle 1, Day 1. All wounds must be fully healed on Cycle 1, Day 1.
* Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease or pulmonary disease
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at screening or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1, Day 1
* History of other malignancy which could affect compliance with the protocol or interpretation of results. Patients with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are allowed. Patients with a malignancy that has been treated with curative intent will also be allowed if the malignancy has been in remission without treatment for >/= years prior to Cycle 1, Day 1.
* Presence of positive test results for Hepatitis B (Hepatitis B surface antigen [HBsAg] and/or total HB core antibody [anti-HB-c]) or Hepatitis C (Hepatitis C virus [HCV] antibody serology testing). Patients positive for anti-HB-c are eligible only if PCR is negative for HBV DNA.
* Known history of HIV seropositive status
* Primary CNS malignancy, or untreated/active CNS metastases
* Pregnancy, lactation or breastfeeding
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Incidence of dose dose limiting toxicities (DLTs) by NCI CTCAE, v4.0 | Days 1-28 of Cycle 1
Nature of dose limiting toxicities (DLTs) by NCI CTCAE, v4.0 | Days 1-28 of Cycle 1

SECONDARY OUTCOMES:
Incidence of adverse events by NCI CTCAE, v4.0 | Up to 1 year
Nature of adverse events by NCI CTCAE, v4.0 | Up to 1 year
Severity of adverse events by NCI CTCAE, v4.0 | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle A. Rooney, M.B., Ch.B., Study Director — Genentech, Inc.
Locations (5):
- United States (5):
  - Scottsdale, Arizona
  - Santa Monica, California
  - Aurora, Colorado
  - Chicago, Illinois
  - Nashville, Tennessee